CLINICAL TRIAL: NCT03696953
Title: The Efficacy of Probiotics to Reduce Antepartum Group B Streptococcus Colonization
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Wake Forest University Health Sciences (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: R21HD095320 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Group B Streptococcus Carrier in Childbirth; Gastrointestinal Symptoms
Keywords: Probiotics; Pregnancy; Group B Streptococcus; Gastrointestinal symptoms

STUDY DESIGN:
Intervention Model Description: Healthy pregnant participants will be randomly assigned to one of two groups (Probiotic vs Placebo) that are blind to participants and researchers. Both groups will take one capsule daily and have the same study measures at the same times.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind Randomized Placebo Controlled Trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Florajen3 Combination Probiotic Product 15 billion CFU per capsule
  1 capsule daily from 28 weeks until the time of birth.
  Interventions: Biological: Florajen3
- Placebo (No Intervention): Microcrystalline Cellulose

INTERVENTIONS:
Biological: Florajen3 — Probiotic combination product One capsule daily by mouth.
  Arms: Probiotic

SUMMARY:
This study is a randomized double blind, placebo controlled trial to determine the efficacy of an oral probiotic in reducing antenatal Group B Streptococcus colonization. The goal of this study is to demonstrate that women in the probiotics group will experience; (1) reduced GBS prenatal colonization at 36± 2 weeks gestation and lower levels of GBS colonization, (2) less need for intrapartum antibiotic prophylaxis and (3) fewer prenatal gastrointestinal symptoms compared to women in the placebo group.

Intrapartum measures were added and IRB approved in Feb 2020 as a pilot and feasibility substudy. The goals of this study are as follows: (1) Explore the effect of antepartum exposure to Florajen3 on maternal and neonatal residual GBS and the maternal microbiome. We anticipate that (1)At the time of labor, more women in the probiotics group will test negative for GBS on vaginal to rectal swabs compared to those in the placebo group and (2) Fewer neonates born to women in the probiotic group will have GBS on nasal-oral pharynx cultures within several hours of birth compared to those born to neonates in the control group.

DETAILED DESCRIPTION:
Group B streptococcus (GBS) is the most prevalent cause of perinatal infection, with mortality and profound comorbidities for neonates. Vaginal and gastrointestinal (GI) colonization with GBS occurs in up to 30% of adult women, with highest rates in African Americans. Pregnant women can pass GBS to their fetuses during vaginal birth, putting them at risk for Early Onset Group B Streptococcus Disease (EOGBSD), which is associated with a neonatal mortality rate of 5-10% and morbidity of approximately 50%. The Centers for Disease Control and Prevention (CDC) 2010 guidelines require universal antepartum GBS screening by vaginal to rectal cultures of all women at 35-37 weeks gestation, and intravenously administered intrapartum antibiotic prophylaxis (IAP) of two or more doses if a woman is found to be colonized with GBS. While use of these guidelines has significantly reduced EOGBSD incidence from 1.7 per 1,000 live births to 0.34-0.37, up to 30% of laboring women and their fetuses are exposed to IAP. Complications associated with IAP are significant for both the mother (increased incidence of antibiotic resistance, allergic sensitization, diarrhea including Clostridium difficile, and fungal infections) and neonate (gut dysbiosis, opportunistic infections, and allergic risk). The proposed study will test a low-cost, safe, innovative approach to reduce prenatal colonization with GBS, while adhering to CDC guidelines for EOGBSD prevention. Investigators hypothesize that women who ingest a commercially available oral probiotic combination product (Florajen3, containing Lactobacillus acidophilus, Bifidobacterium lactis, and Bifidobacterium longum) daily from 28 weeks gestation through the time of labor will have a lower risk of GBS colonization compared to women taking placebo. The purpose of this Phase 2 placebo-controlled, double blind, randomized controlled trial (RCT) is to determine the efficacy of once daily ingestion of Florajen3 by healthy low-risk pregnant women from 28 weeks gestation until the time of labor to (a) reduce the proportion of women with GBS colonization and thus (b) reduce the number of women who receive IAP. Investigators expect this intervention to alter the vaginal and rectal microbiota by (c) increasing Lactobacillus colony counts, (d) decreasing GBS colony counts, and (e) reducing GI symptoms. In preparation for this RCT, the research team conducted two preliminary studies (one in vitro, one in vivo), an integrative review of the literature regarding the use of prenatal probiotics, and a systematic review on probiotics and urogynecologic infections. The literature and preliminary work support the safety, tolerability, and potentially high impact of the oral probiotic as an innovative, low-risk, easy-to-use intervention to reduce GBS colonization during pregnancy and significantly reduce exposure of mothers and infants to IAP and the associated complications. If positive, findings from this study will shift the paradigm in clinical practice and be used to design and conduct a larger RCT to extend the science of nursing, midwifery, obstetrics, microbiology, clinical nutrition, and infectious disease for care of pregnant women and their infants.

Approximately 10% of women who tested negative for GBS at 36 weeks will become positive at the time of labor and birth. This "residual GBS" may be responsible for cases of EOGBSD cases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (≥ 18 years of age) pregnant women who are 28±2 weeks gestation at enrollment [calculated from the first day of Last Normal Menstrual Period (LNMP) and/or ultrasound (US)]
* With: No obstetric complication* (e.g., pre-eclampsia, gestational diabetes, multiple gestation)
* No fetal complication (e.g., birth defect, intrauterine growth restriction)
* No medical complication (e.g., hypertension, diabetes mellitus)
* Who do not currently ingest an over the counter probiotic supplement (not including yogurt)
* Who can both speak and read English
* Who regularly attend prenatal care (defined as not > 1 prior missed appointment during this pregnancy)
* No Hypersensitivity reaction to β-lactam antibiotics

Exclusion Criteria:

* Those less than 18 years of age
* Non-pregnant women
* Later in pregnancy than 30 weeks gestation at enrollment [per LNMP and/or US]
* Those with an obstetric, fetal or medical complication of pregnancy
* Pregnant women who have a history of GBS bacteriuria during the current pregnancy or have previously given birth to a GBS affected child
* Women who are currently ingesting an over the counter probiotic supplement (except for yogurt)
* Women who are planning an elective repeat cesarean birth
* Women who do not speak and read English
* Women with a history of missing more than one scheduled prenatal visit during this pregnancy
* Hypersensitivity reaction to β-lactam antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 109 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Hanson, PhD, Principal Investigator — Marquette University, College of Nursing
Locations (1):
- Aurora Sinai Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanson L, Vandevusse L, Duster M, Warrack S, Safdar N. Feasibility of oral prenatal probiotics against maternal group B Streptococcus vaginal and rectal colonization. J Obstet Gynecol Neonatal Nurs. 2014 May-Jun;43(3):294-304. doi: 10.1111/1552-6909.12308. Epub 2014 Apr 22. PMID 24754328
- [Background] Hanson L, VandeVusse L, Jerme M, Abad CL, Safdar N. Probiotics for Treatment and Prevention of Urogenital Infections in Women: A Systematic Review. J Midwifery Womens Health. 2016 May;61(3):339-55. doi: 10.1111/jmwh.12472. PMID 27218592
- [Background] VandeVusse L, Hanson L, Safdar N. Perinatal outcomes of prenatal probiotic and prebiotic administration: an integrative review. J Perinat Neonatal Nurs. 2013 Oct-Dec;27(4):288-301; quiz E1-2. doi: 10.1097/JPN.0b013e3182a1e15d. PMID 24164813
- [Background] Hanson L, Vandevusse L. Probiotics are food; herbs are plants; what's the risk? Informed consent for complementary and integrative therapies. J Perinat Neonatal Nurs. 2010 Jul-Sep;24(3):201-4. doi: 10.1097/JPN.0b013e3181e8f930. No abstract available. PMID 20697235
- [Background] Dunn AB, Hanson L, VandeVusse L, Leslie S. Through the Microbial Looking Glass: Premature Labor, Preeclampsia, and Gestational Diabetes: A Scoping Review. J Perinat Neonatal Nurs. 2019 Jan/Mar;33(1):35-51. doi: 10.1097/JPN.0000000000000375. PMID 30676461
- [Background] Simonson J, Haglund K, Weber E, Fial A, Hanson L. Probiotics for the Management of Infantile Colic: A Systematic Review. MCN Am J Matern Child Nurs. 2021 Mar-Apr 01;46(2):88-96. doi: 10.1097/NMC.0000000000000691. PMID 33315632
- [Background] Malloy E, Kates A, Watson L, VandeVusse L, Safdar N, Hanson L. Laboratory Analysis Techniques for the Perinatal Microbiome: Implications for Studies of Probiotic Interventions. J Perinat Neonatal Nurs. 2020 Jul/Sep;34(3):239-250. doi: 10.1097/JPN.0000000000000496. PMID 32697544
- [Result] Hanson L, VandeVusse L, Forgie M, Malloy E, Singh M, Scherer M, Kleber D, Dixon J, Hryckowian AJ, Safdar N. A randomized controlled trial of an oral probiotic to reduce antepartum group B Streptococcus colonization and gastrointestinal symptoms. Am J Obstet Gynecol MFM. 2023 Jan;5(1):100748. doi: 10.1016/j.ajogmf.2022.100748. Epub 2022 Sep 13. PMID 36108911
- [Derived] Hanson L, Albert K, Malloy E, Singh M, Kallay M, Brandt A, Morris C, Kleber D, Forgie M. Participant Personal Characteristics and Adherence to Oral Capsules: A Secondary Analysis of a Randomized Placebo-Controlled Trial of Antenatal Probiotics. J Midwifery Womens Health. 2025 May-Jun;70(3):452-459. doi: 10.1111/jmwh.13686. Epub 2024 Oct 1. PMID 39351987

RESULTS

PARTICIPANT FLOW:
Groups:
- Probiotic: Florajen3 Combination Probiotic Product 15 billion CFU per capsule
  1 capsule daily from 28 weeks until the time of birth.
  Florajen3: Probiotic combination product One capsule daily by mouth.
Period: Overall Study
Arm/Group | Probiotic | Placebo
Started | 55 | 54
Completed | 39 | 44
Not Completed | 16 | 10
Not completed — Withdrawal by Subject | 6 | 1
Not completed — missed GBS swabs | 2 | 2
Not completed — lost study bottle containing capsules | 2 | 0
Not completed — Premature birth | 1 | 4
Not completed — Gestational hypertension | 1 | 1
Not completed — Gestational diabetes | 2 | 1
Not completed — Fetal demise-Genetic abnormality | 1 | 0
Not completed — Changed prenatal provider | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic | Placebo | Total
Number analyzed (Participants) | 39 | 44 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (5.4) | 28.4 (5.5) | 28.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 44 | 83
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 16 | 33
  White | 19 | 23 | 42
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Parity [Count of Participants; unit: Participants]
  Nulliparous | 16 | 20 | 36
  Multiparous | 23 | 23 | 46
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Qualitative GBS Culture Result
Description: Qualitative GBS culture results
Time Frame: 36 weeks gestation
Population: Number of GBS Culture Positive Participants at 36 week standard of care cultures
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 39 | 44
Participants
  Positive GBS culture | 6 | 9
  Negative GBS culture | 33 | 35
Statistical Analysis 1: Comparison: Probiotic; Test type: Other — t test comparing; p = 0.05, t-test, 2 sided

2. Secondary Outcome: GBS Quantitative Colony Counts in Colony Forming Units (CFU)
Description: Amount of GBS on each vaginal and rectal swab. Each swab was vortexed in 1 mL of PBS and plated onto Granada agar. Quantitative GBS colonization measured as the number of GBS colonies on Granada agar plate multiplied by the inverse of the dilution factor. The results were reported in CFU. No GBS present indicates negative. Positive results are reports numerically.
Time Frame: 36 weeks gestation
Population: Mean GBS Colony Forming Units (CFU)
Measure: Mean (Standard Deviation); unit: CFU
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 39 | 44
CFU
  Vaginal | 11.32 (6.65) | 317.1 (1957.1)
  Rectal | 604.2 (2684.2) | 2046.6 (12805.4)
Statistical Analysis 1: Comparison: Probiotic vs Placebo; Test type: Other; p = 0.73, t-test, 2 sided
Statistical Analysis 2: Comparison: Probiotic vs Placebo; Test type: Other — T test; p = 0.05, t-test, 2 sided

3. Secondary Outcome: Antepartum Gastrointestinal Symptom Assessment
Description: Antepartum Gastrointestinal Symptom Assessment Scores
  The Antepartum Gastrointestinal Symptom Assessment is a composite of 10 GI symptoms (Nausea, Vomiting, Diarrhea, Sour Taste, Bad Breath, Burping/Belching, Bloating, Heartburn, Diarrhea, Constipation) each scored from 1 (no problem) to 5 (very severe problem), leading to a composite score between 10-50. Lower scores indicate fewer and/or less severe GI symptoms. Higher scores indicate more frequent and/or more severe GI symptoms.
Time Frame: 36 weeks gestation
Population: The Antepartum Gastrointestinal Symptom Assessment is a composite of 10 GI symptoms (Nausea, Vomiting, Diarrhea, Sour Taste, Bad Breath, Burping/Belching, Bloating, Heartburn, Diarrhea, Constipation) each scored from 1 (no problem) to 5 (very severe problem), leading to a composite score Minimum of 10 and maximum of 50. Lower scores indicate fewer and/or less severe GI symptoms. Higher scores indicate more frequent and/or more severe GI symptoms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 39 | 44
score on a scale
  Baseline (28 week) AP-GI-SA Score | 14.7 (3.2) | 16.2 (4.8)
  36 week AP-GI-SA Score | 13.58 (2.77) | 15.64 (3.96)
Statistical Analysis 1: Comparison: Probiotic vs Placebo; Comparison of 36 week AP-GI-SA Scores between probiotic and placebo groups at 36 weeks; Test type: Other — T test; p = 0.01, t-test, 2 sided

4. Other Pre Specified Outcome: Intrapartum GBS Culture Result
Description: Number of women with positive GBS vaginal to rectal colonization at the time of admission to the hospital for labor and birth. This measure was only collected on participants in the substudy.
Time Frame: At the time of admission to the hospital for labor and birth (intrapartum) (Time frame will vary by participant and their health status, at or beyond 36 weeks 0/7 days gestation until 42 weeks 0/7 days gestation)
Population: Qualitative GBS culture positive or negative. No GBS on the plate indicates a negative culture. Any GBS on the plate indicates a positive culture.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 14 | 16
Participants
  Intrapartum Culture Positive | 3 | 3
  Intrapartum Culture Negative | 11 | 12
  GBS culture changed to Positive (36 weeks to negative Intrapartum | 1 | 2
  GBS culture changed to Negative (36 weeks to positive Intrapartum | 1 | 0
Statistical Analysis 1: Comparison: Probiotic vs Placebo; Test type: Other — T test; p = 0.05, t-test, 2 sided

5. Other Pre Specified Outcome: Neonatal GBS Oral/Nasopharynx Colonization
Description: Number of Neonates with Positive GBS ) oral/nasopharynx colonization within 1-2 hours of life
Time Frame: 1-2 hours of life
Population: Neonatal oral/nasopharynx swabs. No GBS on plate indicates a negative culture. Any GBS present indicates a positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 14 | 16
Participants | 0 | 0
Statistical Analysis 1: Comparison: Probiotic vs Placebo; Test type: Other — T test; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From 28 weeks gestation (baseline/enrollment) to 2 months post birth
Arm/Group | Probiotic | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03696953/Prot_SAP_002.pdf
  • Informed Consent Form (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03696953/ICF_003.pdf